CLINICAL TRIAL: NCT03718858
Title: Evaluating the Impact of Interscalene Brachial Plexus Block on Sleep-disordered Breathing in Patients Undergoing Ambulatory Shoulder Surgery. A Two-arm, Prospective, Parallel, Double Blind Randomized -Controlled Trial
Brief Title: The Impact of Interscalene Block on Sleep Disordered Breathing
Acronym: OSA-ISB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018-0037-B
Record Dates: First submitted 2018-09-10; First posted 2018-10-25 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
Keywords: sleep; Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Intervention Model Description: This is two-arm, prospective, parallel, double blind, multi center, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: On the day of surgery, patients will be randomly assigned (1:1) to one of two groups according to a computer-generated list. The patients, the clinical care team (anesthesiologist providing intraoperative care, nurses, and surgeons), data collectors, outcome adjudicators, and the study statisticians will all remain blinded to randomization and group allocation. The anesthesiologist who will perform the intervention will be aware of group allocation, but the anesthesiologist providing intraoperative care will remain blinded. Situations such as patient refusal at any time of the study, any adverse event or complication necessitating withholding the intervention would result in voluntary un-blinding of study investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block (Experimental): Under sterile precautions, a high frequency linear array transducer [6-13 Megahertz (MHz), Sonosite M-Turbo] probe will be placed in the transverse plane over the interscalene groove to visualize the carotid artery and the C5 and C6 nerve roots of the brachial plexus between the anterior and middle scalene muscles. A 5 cm 22 G insulated needle will then be inserted in line with the US probe in a lateral-to-medial approach until the needle tip is adjacent to the C5 and C6 roots. After negative aspiration for blood, 15 mL ropivacaine 0.5% will be injected in 5 mL aliquots in order to achieve spread adjacent to C5 and C6 nerve roots.
  Interventions: Procedure: Interscalene Block
- Superior Trunk Nerve block (Active Comparator): Under sterile precautions, a high frequency linear array transducer [6-13 Megahertz (MHz), Sonosite M-Turbo] probe will be placed in the transverse plane over the interscalene groove to visualize the carotid artery and the C5 and C6 nerve roots of the brachial plexus between the anterior and middle scalene muscles. The superior trunk will be identified by tracing the C5 and C6 nerve roots caudally towards the supraclavicular fossa on the anterior lateral portion of the neck. A 5 cm 22 G insulated needle will then be inserted in line with the US probe in a lateral-to-medial approach until the needle tip is properly positioned. After negative aspiration for blood, 15 mL ropivacaine 0.5% will be injected in 5 mL aliquots.
  Interventions: Procedure: Superior Trunk Nerve Block

INTERVENTIONS:
Procedure: Interscalene Block — 15 mL ropivacaine 0.5% will be injected in 5 mL aliquots in order to achieve spread adjacent to C5 and C6 nerve roots.
  Arms: Interscalene block
Procedure: Superior Trunk Nerve Block — 15 mL ropivacaine 0.5% will be injected in 5 mL aliquots in order to achieve spread adjacent to Superior Trunk Nerve.
  Arms: Superior Trunk Nerve block

SUMMARY:
This is a randomized controlled trial evaluating the impact of interscalene block on worsening of upper airway collapse in sleep disordered breathing for patients undergoing ambulatory shoulder surgery.

DETAILED DESCRIPTION:
Sleep disordered Breathing (SDB), closely associated with obesity, is a highly prevalent, serious, and often unrecognized breathing disorder resulting from repeated upper airway collapse, decreased oxygen levels, and a very high risk of life threatening complications at the time of surgery. Current guidelines recommend using regional as opposed to general anesthesia in SDB patients to minimize risks and the use of strong narcotic medications. It is unclear whether interscalene block in use for analgesia (pain relief) may actually worsen the severity of SDB by invariably freezing the phrenic nerve, thereby temporarily paralyzing the diaphragm.

This novel clinical trial will examine whether or not ISB increases the rate of upper airway obstruction or collapse during sleep and other dangerous postoperative complications seen in patients with SDB following shoulder surgeries.

The Primary Objective of the study is to evaluate the impact of ISB on the oxygen desaturation index (sleep apnea severity) in untreated SDB patients undergoing ambulatory shoulder surgery compared to patients who do not receive ISB.

Secondary Objectives are: 1) To evaluate the impact of hemidiaphragmatic paresis on impairment in pulmonary function; 2) To evaluate the impact of impairment in pulmonary function on the oxygen desaturation index (ODI); 3) To assess the incidence of important perioperative clinical outcomes such as hypoxemia, recurrent respiratory events, delayed discharge, and resource utilization in SDB patients undergoing ambulatory shoulder surgery compared to patients who do not receive ISB; and 4) To assess important analgesia related outcomes such as: time to onset of pain, intraoperative and postoperative opioid consumption, hourly and daily VAS pain scores, opioid related side effects, patient satisfaction with analgesia, and presence/absence of nerve block complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ( >18 to 80 years);
* American Society of Anesthesiology (ASA) physical status I-IV;
* Undergoing elective ambulatory shoulder surgery such as shoulder replacement, acromioplasty, rotator cuff repair, or Bankart procedure under general anesthesia.

Exclusion Criteria:

* Past history of head, neck or thoracic surgery (e.g., OSA corrective surgery);
* Pregnancy or lactation;
* Phrenic nerve stimulators;
* Local anesthetic allergy;
* Previous diaphragmatic paralysis;
* Inability to communicate with health care providers or the research personnel, inability to perform breathing maneuvers such as spirometry, or inability to follow instructions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen desaturation index (ODI) from baseline to the night of surgery (post- operation) (N1). | Time of measurements will be at baseline (pre operatively) and within 24 hours post-operatively (night of surgery)
  All patients will undergo a portable overnight oximetry study at home to establish the baseline oxygen saturation measured hourly. Oxygen Desaturation Index (ODI), which is defined as a 4% drop in oxygenation from the baseline, and calculated as events occurring per hour during the recording time; the minimum and mean oxygen saturation ; and the cumulative total of recoded time below an oxygen saturation of 90%, CT90). Patients with preoperative ODI with more than a score of 10 will be considered at risk of SDB. A change from baseline will be examined and compared between the two groups.

SECONDARY OUTCOMES:
Change in amplitude of diaphragmatic excursion with breathing maneuvers, between before and after surgery (measured by ultrasound) | Time of measurements will be within 1 hour before surgery, and within 1 hour after surgery. It will take around 10-15 minutes.
  Rate of diaphragmatic function (complete, partial, or none) will be assessed before and after surgery using M-Mode Ultrasound. Assessment will be performed during quiet breathing, sniffing, and deep breathing. After surgery diaphragmatic paresis will be indicated by a flat trace (absence of excursion) with quiet and deep breathing and/or with paradoxical motion. Measurement of amplitude of excursion will be made when partial paresis is observed. Using the sniff maneuver, complete hemi-diaphragmatic paresis (reduction of >75% from baseline) and partial paresis (reduction of 25-75%from baseline) will be recorded. Rate will be assessed in the basal state (i.e. before regional anesthesia) to establish a baseline, and again in the post-operative period.
Change in pulmonary function before and after surgery, as measured by bedside spirometry | Time of measurements will be within 1 hour before surgery, and within 1 hour after surgery. It will take around 5-10 minutes.
  Change in pulmonary function tests [Forced vital capacity (FVC), forced expiratory volume in 1s (FEV1), Expiratory reserve volume (ERV) and peak expiratory flow (PEF) ], between before and after surgery will be measured by bedside spirometry
Post operative respiratory events | Within 24 hours of the time of surgery
  Respiratory events in recovery room (Oxygen saturation < 90% (3 episodes), bradypnea < 8 breaths / min (3 episodes), apnea ≥ 10s (1 episode) will be recorded.
Visual Analogue Scale (VAS) pain scores | 8 hours and 24 hours after surgery.
  Measurement of hourly and daily Visual Analogue Scale (VAS) pain scores. VAS: 10cm scale where 0=no pain, 10=worst pain.
Analgesia requirements | Day 1 of surgery.
  Opioid and other pain killers consumption will be recorded intra and post-operatively
Patient satisfaction with analgesia | 8 hours and 24 hours after surgery.
  A follow up call will be made on day 1 and day 30 to collect overall satisfaction with pain control. Overall satisfaction will be assessed on a 7-point Likert scale of 1-not at all satisfied with pain control, 2-mostly unsatisfied with pain control, 3-slightly unsatisfied with pain control, 4-no opinion, 5-slightly satisfied with pain control, 6-mostly satisfied with pain control, 7-completely satisfied with pain control

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mandeep Singh, Principal Investigator — Women's College Hospital and Toronto Western Hospital, University Health Network; Dr. Richard Brull, Principal Investigator — Women's College Hospital and Toronto Western Hospital, University Health Network
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, ON Ontario
  - Toronto Western Hospital, Toronto, Ontario